CLINICAL TRIAL: NCT00616447
Title: A 12-week, Double-blind, Randomized, Placebo-controlled Multicentered Study Evaluating Efficacy and Safety of High-frequency Repetitive Transcranial Magnetic Stimulation (rTMS) Treatment in Patients With Generalized Anxiety Disorder (GAD)
Brief Title: rTMS Treatment in Patients With General Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Military Medical Academy, Bulgaria (Other)
Responsible Party: Principal Investigator, Dr. Roumen Milev, Professor of Psychiatry and Psychology, Head, Department of Psychiatry Queen's University, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PSIY-270-07
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Device: Repetitive transcranial magnetic stimulation
- 2 (Sham Comparator)
  Interventions: Device: placebo sham

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — 6 weeks of repetitive transcranial magnetic stimulation . Treatment comprises of stimulation with rTMS frequency 20Hz, intensity 110% of MT, 20 trains, 9 sec/train, 51 sec ITI applied over right dorsolateral prefrontal cortex by a figure eight shaped coil. Treatment will be given 5 times a week for 4 weeks, 3 times a week during Week 5 and 2 times a week during Week 6.
  Other Names: rTMS machine (MagPro, Medtronic).
  Arms: 1
Device: placebo sham — Sham treatment will mimic active treatment mentioned above.
  Other Names: rTMS machine (MagPro, Medtronic).
  Arms: 2

SUMMARY:
This study will compare the change detected by a standardized rating scale (Hamilton Anxiety Rating Scale) scores in the active treatment group as compared to sham (placebo) group after 6 weeks of rTMS treatments. It is hoped that 6 weeks of rTMS treatment will lead to improvement of core symptoms in patients with GAD.

ELIGIBILITY:
Inclusion Criteria:

* signed patient informed consent;
* primary GAD diagnosis;
* HARS >=15;
* male/female 18-65 years;
* without GAD pharmacotherapy at least last 2 weeks or if they are taking GAD medication it must be stable for at least 6 weeks prior to the start of the study and not be changed during the 6 weeks of the study treatment phase.
* Individual or group supportive psychotherapy may continue during the study but will not be allowed to start new psychotherapy during the 6 weeks of the study treatment phase.

Exclusion Criteria:

* current serious Axis I schizophrenia, bipolar I, MDD;
* other primary Axis I in the opinion of investigator;
* HDRS >=18;
* metallic implant in cranium except mouth;
* severe/unstable medical conditions;
* ect within last 3 months;
* history epilepsy;
* neurological disorder leading to increased intracranial pressure;
* severe cardiac disorder/intracardiac lines/pacemakers;
* current suicide risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Hamilton Anxiety Rating Scale (ham-a) | baseline, week 2, 4, 6, 8, 12

SECONDARY OUTCOMES:
Clinical Global Impression | baseline, 2, 4, 6, 8, 12
Hamilton Depression Rating Scale-21 | baseline, week 2, 4, 6, 8, 12
Pittsburgh Sleep Quality Index | baseline, week 2, 4, 6, 8, 12
SF-36 QOL version (1) | baseline, week 2, 4, 6, 8, 12
Visual Analogue Scales | baseline, week 2, 4, 6, 8, 12

CONTACTS AND LOCATIONS:
Overall Officials: Roumen Milev, MD, Study Chair — Queen's University
Locations (2):
- Military Medical Academy, Sofia, Bulgaria
- Providence Care Mental Health Services, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Dilkov D, Hawken ER, Kaludiev E, Milev R. Repetitive transcranial magnetic stimulation of the right dorsal lateral prefrontal cortex in the treatment of generalized anxiety disorder: A randomized, double-blind sham controlled clinical trial. Prog Neuropsychopharmacol Biol Psychiatry. 2017 Aug 1;78:61-65. doi: 10.1016/j.pnpbp.2017.05.018. Epub 2017 May 19. PMID 28533148